CLINICAL TRIAL: NCT00611117
Title: Mechanisms of the Effect of Physical Activity on the Adaptation to a High-Fat Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PBRC 27017; 58-6535-5-071
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2016-01

CONDITIONS: Healthy
Keywords: adaptation to high fat diet; activity; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): High intensity exercise and high fat diet
  Interventions: Other: Physical Activity Level
- 2 (Experimental): Low intensity exercise and high fat diet
  Interventions: Other: Physical Activity Level

INTERVENTIONS:
Other: Physical Activity Level — High vs. low physical activity during a high fat diet consumption.

SUMMARY:
The study is designed to determine the effect of high physical activity level vs. low physical activity level on the adaptation to a high fat diet.

DETAILED DESCRIPTION:
A high fat diet is linked to weight gain and obesity. An adjustment to the acute exposure to high fat diet is not abrupt and takes time. In a previous study from our laboratory, it has been shown that high level of physical activity can accelerate the adaptation to a high fat diet by increasing fat oxidation. In this study we will determine the mechanism involved in this adjustment. Our hypotheses are:

1. High fat diets decrease skeletal muscle glucose metabolism and decrease mitochondrial biogenesis through the upregulation of PDK4 and downregulation of PGC1α; increased physical activity will prevent these deleterious effects.
2. A high fat diet will increase hepatic and skeletal muscle lipid; increased physical activity will prevent these deleterious effects.
3. These effects are more pronounced in individuals with a low mitochondrial content

ELIGIBILITY:
Inclusion Criteria:

* Both genders and all races will be invited to participate
* BMI > 19 and < 35 kg/m2
* Age 18-35
* Women will be asked to participate in the follicular phase of the menstrual cycle as determined by menstrual history and a negative pregnancy test will be recorded prior to participation
* Willing and able to walk on a treadmill at a pace of 3 mph at 3%grade for 3-4 hours/day for 3 consecutive days
* Willing to eat only and all foods provided by Pennington for 9 days on 2 occasions (18 days)
* Willing to stop alcohol consumption for the duration of the study
* Able come to Pennington for meals and tests for 20 days 12 of these inpatient.

Exclusion Criteria:

* Significant renal, hepatic, endocrine, pulmonary, cardiac or hematological disease (for the consent form you will have to use kidney, liver, etc )
* You abuse alcohol or illegal drugs or are unable to avoid alcohol or caffeine prior to testing
* Smokers
* Unable or unlikely to eat all and only food provided by the PBRC metabolic kitchen.
* Pregnant or planning to become pregnant
* Corticosteroid use in previous two months
* Chronic use of anti-diabetic, anti-hypertensive, or other medications known to affect fat metabolism
* Use of Depo-Provera, hormone implants or estrogen replacement therapy
* Irregular menstrual cycles
* Post-menopausal women
* Weight gain or loss of > 3kg in the last 6 months
* Unable or unwilling to perform treadmill walking at the required speed and incline to achieve 1.8*RMR
* History or family history of blood clots deep vein thrombosis or pulmonary embolism)
* Poor circulation, bypass operation on legs, blood coagulation disorders, diagnosed peripheral arterial or vascular disease, cramping pain in your muscle during exercise or nerve damage in your legs.
* You had major surgery on the abdomen, pelvis or legs within previous 3 months.
* You have cancer
* You have rheumatoid disease/ walking or joint problems
* You are claustrophobic
* You are depressed or have an eating disorder
* You demonstrate a style of interpersonal relationships that would inhibit successful completion of the study

For the MRS / MRI, the following exclusion criteria apply:

* Individuals who have a heart pacemaker, defibrillator, or non-removable hearing aid
* Individuals with any clips or metal plates in their head
* Individuals who have any artificial limbs or prosthetic devices
* Individuals who were ever injured by a metallic foreign body which was not removed
* Individuals with bridgework held in place by magnets

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
To determine the effects of a high fat diet [at both low and high physical activity] on • Sk muscle PGC1α and PDK4 mRNA and protein • Glucose oxidation • Fatty acid oxidation • Hepatic and skeletal muscle lipid • VO2 max • Mitochondr | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Smith, Principal Investigator — Pennington Biomedical Research Center; George Bray, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States